CLINICAL TRIAL: NCT00026650
Title: Evaluation of Late Effects and Natural History of Disease in Patients Treated With Radiotherapy
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000074; 00-C-0074; NCT00436813 (obsolete NCT alias)
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12-16

CONDITIONS: Cancer
Keywords: Late Effects; Radiation Therapy; Cancer; Natural History
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Cohort 1: Patients who have received radiotherapy in the ROB and may or may not be officially entered on a clinical protocol.

SUMMARY:
BACKGROUND

* This protocol acknowledges that it is in the interest of the NIH and ROB, as well as our participants, to continue to follow those who have been treated with radiotherapy at ROB and are not otherwise eligible for current active research protocols.
* It also provides a mechanism for the correlation and interpretation of disparate data for research into the long term side effects and outcomes for a variety of disease entities and treatments, such as combined modality treatment, MoAb, PDT, radiation modifiers,

intraoperative radiotherapy, etc.

OBJECTIVE

-The primary objective of this protocol is to assess the late effects of treatment and the natural history of disease through collection of data from any standard procedures performed as part of follow up care on participants previously treated with radiotherapy.

ELIGIBILITY

-Participants who received radiation therapy.

DESIGN

* This is a natural history protocol in which long-term follow up data will be collected from participants who received radiation therapy.
* It will be made clear to participants in the consent form, that data collected during their follow-up may be used anonymously for publications concerning the natural history of disease processes and long-term effects of treatment.

DETAILED DESCRIPTION:
BACKGROUND

* This protocol acknowledges that it is in the interest of the NIH and ROB, as well as our participants, to continue to follow those who have been treated with radiotherapy at ROB and are not otherwise eligible for current active research protocols.
* It also provides a mechanism for the correlation and interpretation of disparate data for research into the long term side effects and outcomes for a variety of disease entities and treatments, such as combined modality treatment, MoAb, PDT, radiation modifiers,

intraoperative radiotherapy, etc.

OBJECTIVE

-The primary objective of this protocol is to assess the late effects of treatment and the natural history of disease through collection of data from any standard procedures performed as part of follow up care on participants previously treated with radiotherapy.

ELIGIBILITY

-Participants who received radiation therapy.

DESIGN

* This is a natural history protocol in which long-term follow up data will be collected from participants who received radiation therapy.
* It will be made clear to participants in the consent form, that data collected during their follow-up may be used anonymously for publications concerning the natural history of disease processes and long-term effects of treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

ROB investigator deems that it is in the best interests of the participant and the NCI/ROB for the participant to be seen in follow-up in the ROB clinic.

Participant is able to provide informed consent.

Participant must have a primary physician in the community to whom records and appropriate follow-up management can be given. Social services will be enlisted for any participants who lack health insurance, etc.

Participants who have received radiotherapy.

Age greater than or equal to 18 years of age

EXCLUSION CRITERIA:

Participants who are on an interventional research protocol at NIH at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received radiation
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2000-02-14 (Actual)

PRIMARY OUTCOMES:
Assessment of the late effects of treatment and the natural history of disease | Ongoing
  Description of late effects of radiation treatment and the natural history of diseases being studied.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2000-C-0074.html